CLINICAL TRIAL: NCT06550102
Title: Drug Response Profiling (DRP) Registry Zurich for Hematological Malignancies
Acronym: DRP_ZH
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02189
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hematological Malignancies
Keywords: registry; DRP; acute lymphoblastic leukemia; blood cancer
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematological malignancy: Patients witha diagnosis of hematological malignancy (primary, relapsed or refractory) including leukemia, myeloma or lymphoma

SUMMARY:
This study is a prospective, non-randomized feasibility study of drug response profiling (DRP) in pediatric blood cancers. Primary cancer cells are isolated from patients and screened ex vivo at single-cell resolution using automated fluorescence microscopy. Drug sensitivity fingerprints are integrated with genetic annotations to inform the treating physician about personalized treatment options. The study aims to determine the practicability of real-time drug response profiling and its actionability in identifying patient-specific cancer dependencies in refractory disease settings.

DETAILED DESCRIPTION:
This observational study offers a platform to assess the drug sensitivity of primary leukemia cells ex vivo. The cancer cells are co-cultured in multi-well plates with supporting mesenchymal stroma cells and exposed to a library of both conventional (e.g. steroids, vincristine, asparaginase) as well as targeted chemotherapeutic agents (e.g. tyrosine kinase inhibitors, proteasome inhibitors, B-cell lymphoma 2 (BCL2) inhibitors). Cells are imaged in parallel by high-content microscopy and subsequently segmented and classified by morphology and surface antigen expression. Cell viability is quantified relative to dimethyl sulfoxide (DMSO) and as a function of drug concentration. From the measured cell counts drug-specific sensitivity parameters (e.g. half-maximal inhibitory concentration IC50, maximal inhibition Imax, area under the curve AUC) and their z-scores across the patient cohorts are calculated. Drug response profiles are correlated to clinical response after a steroid pre-phase at day 8 and multiple minimal residual disease (MRD) timepoints measured by flow cytometry (FCM) or polymerase chain reaction (PCR) as defined by the trial protocol. Data on clinical response to treatment and outcome will be enquired from the treating physician. These include the disease stage (initial diagnosis, 1st relapse, 2nd relapse) and time point of sample collection, the clinical trial and treatment arm the patient is enrolled in and/or any individualized drug treatments. Functional profiling data will be integrated with information about genetic lesions (e.g. tumor protein TP53), subtype-defining translocations such as the Philadelphia chromosome t(9;22)(q34;q11) and surface antigen expression (e.g. clusters of differentiation CD7/19/22/33/117). Cytogenetics and molecular profiling data are collected from the treating clinics in collaboration with the international relapsed acute lymphoblastic leukemia (IntReALL) study group and the international Berlin-Frankfurt-Münster (IBFM) network.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients below the age of 40 years
* Diagnosis of hematological malignancy (primary, relapsed or refractory) including leukemia, myeloma or lymphoma
* Tumor material collected as part of routine diagnostics and willingness to donate tumor material for translational research
* Patient and/or guardian has signed the informed consent of the DRP registry or of a clinical trial which includes DRP as add-on research.

Exclusion Criteria:

* Missing informed consent for the registry or of a clinical trial which includes DRP as add-on research

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and adult patients with hematological malignancies who have undergone bone marrow aspiration, peripheral blood or lymph node biopsies as part of routine diagnostics.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of real-time ex vivo drug screening | 10 days
  Rate of successful single-cell, image-based drug response profiling assays which are reported to the treating physician.

SECONDARY OUTCOMES:
Translation to clinic | 10 day
  Percentage of DRP assays translated into the clinic, i.e. the referring physician decides to treat the patient with one or more of the top-ranking drugs identified by DRP
In vitro sensitivity of cancer cells to drug perturbations | 1 month
  Exploring drug sensitivity and resistance patterns by ex vivo DRP and correlations to genetic characteristics and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Bourquin, MD, PhD, Study Chair — University Children's Hospital Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Frismantas V, Dobay MP, Rinaldi A, Tchinda J, Dunn SH, Kunz J, Richter-Pechanska P, Marovca B, Pail O, Jenni S, Diaz-Flores E, Chang BH, Brown TJ, Collins RH, Uhrig S, Balasubramanian GP, Bandapalli OR, Higi S, Eugster S, Voegeli P, Delorenzi M, Cario G, Loh ML, Schrappe M, Stanulla M, Kulozik AE, Muckenthaler MU, Saha V, Irving JA, Meisel R, Radimerski T, Von Stackelberg A, Eckert C, Tyner JW, Horvath P, Bornhauser BC, Bourquin JP. Ex vivo drug response profiling detects recurrent sensitivity patterns in drug-resistant acute lymphoblastic leukemia. Blood. 2017 Mar 16;129(11):e26-e37. doi: 10.1182/blood-2016-09-738070. Epub 2017 Jan 25. PMID 28122742